CLINICAL TRIAL: NCT05400317
Title: A Randomized, Double-blinded, Active-controlled, Multicenter Phase 3 Clinical Trial and Open-label, Extension Study to Evaluate the Efficacy and Safety of AD-218 in Patients with Mixed Dyslipidemia
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-218
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-218P3
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator : Test group (Experimental): AD-218
  Interventions: Drug: AD-218
- Active Comparator : Control group (Active Comparator): AD-218A
  Interventions: Drug: AD-218A

INTERVENTIONS:
Drug: AD-218 — PO, Once daily(QD), 12weeks
  Arms: Active Comparator : Test group
Drug: AD-218A — PO, Once daily(QD), 12weeks
  Arms: Active Comparator : Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-218

DETAILED DESCRIPTION:
Condition or disease : Mixed Dyslipidemia Treatment Drug : AD-218, AD-218A, Placebo of AD-218, Placebo of AD-218A

ELIGIBILITY:
Inclusion Criteria:

* A man or woman over 19 years old.
* Sign on ICF prior to study participation

Exclusion Criteria:

* History of Fibromyalgia, Myopathy etc (CK ≥ 2 X ULN)
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent change (%) of non-HDL-C from baseline at week 12 | from baseline at 12 weeks
  non-HDL-C at week 12 compared AD-218 with AD-218A

SECONDARY OUTCOMES:
Percent change (%) of non-HDL-C from baseline at week 4, 8 | from baseline at week 4,8
  non-HDL-C at week 4,8 compared AD-218 with AD-218A
Percent change (%) of Lipid panel from baseline at week 4, 8, 12 | from baseline at week 4, 8, 12
  Lipid panel at week 4, 8, 12 compared AD-218 with AD-218A

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Chang Won, M.D., Ph.D, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Yeongnam University Hospital, Daegu, Nam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No